CLINICAL TRIAL: NCT04930536
Title: A Prospective, Multi-centre, Phase IV Clinical Trial to Assess the Safety and Efficacy of Acalabrutinib Capsules in Indian Adult Patients With Chronic Lymphocytic Leukaemia and Relapsed and Refractory Mantle Cell Lymphoma.
Brief Title: Acalabrutinib Study in Indian Patients With Chronic Lymphocytic Leukaemia & Relapsed and Refractory Mantle Cell Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8220C00022
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Chronic Lymphocytic Leukemia and Relapsed and Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Lymphoma, Mantle-Cell | interventions — acalabrutinib

STUDY DESIGN:
Intervention Model Description: A Prospective, Multicentre, Phase-IV study and Clinical trials with a single arm.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib Capsule (Experimental): Single-arm study
  Interventions: Drug: Acalabrutinib capsule

INTERVENTIONS:
Drug: Acalabrutinib capsule — The recommended dose of Acalabrutinib is 100 mg given per oral (PO) twice daily
  Other Names: Calquence®

SUMMARY:
This study is plan to assess the safety and efficacy of Acalabrutinib in Indian patients with chronic lymphocytic leukaemia (CLL) and relapsed and refractory mantle cell lymphoma (MCL)

DETAILED DESCRIPTION:
A prospective, multi-centre, phase IV clinical trial of Acalabrutinib capsules in Indian adult patients with chronic lymphocytic leukaemia (CLL) and relapsed and refractory mantle cell lymphoma (MCL). As per recommendation from Indian health authority, the current phase-IV study is planned with the aim to assess the safety and efficacy profile of Acalabrutinib in Indian patients with CLL/SLL, and patients with MCL who have received at least one prior therapy. The data obtained from the study will help to understand the safety and efficacy profile of Acalabrutinib in Indian patients. Patients will be monitored throughout the study period for Adverse Events of Acalabrutinib

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all of the following inclusion criteria and none of the exclusion criteria apply:

1. Men and Women aged 18yrs or more. 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1, or 2 3. Able to receive all outpatient treatments, all laboratory monitoring, and all radiologic evaluations.

4. The following laboratory parameters:

1. Absolute neutrophil count (ANC) ≥750 cells/μL or ≥500 cells/μL in patients with documented bone marrow involvement, and independent of growth factor support 07 days before the assessment
2. Platelet count ≥50,000 cells/μL or ≥30,000 cells/μL in patients with documented bone marrow involvement, and without transfusion support 07 days before the assessment
3. Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤2.0 x ULN
4. Total bilirubin ≤1.5 x ULN
5. Estimated creatinine clearance of ≥30 mL/min 5. Refractory disease defined as achieving less than partial response with the most recent treatment within 6 months before study entry 6. Provision of signed, written and dated informed consent prior to any study-specific Procedures 7. The patients of either CLL or MCL:

a. CLL patients: i. Treatment naïve or ≥1 prior systemic therapy for CLL ii. Diagnosis of CD20+ CLL that meets published diagnostic criteria (Hallek et al. 2018) iii. An active disease that meets ≥1 of the following iwCLL 2018 criteria for requiring treatment:

1. Evidence of progressive marrow failure as manifested by the development of, or worsening of, anaemia and/or thrombocytopenia. Cut-off levels of Hb <10 g/dL or platelet counts <100 × 109/L are generally regarded as an indication for treatment. However, in some patients, platelet counts <100 × 109/L may remain stable over a long period; this situation does not automatically require therapeutic intervention.
2. Massive (i.e., ≥6 cm below the left costal margin) or progressive or symptomatic splenomegaly.
3. Massive nodes (i.e., ≥10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.
4. Progressive lymphocytosis with an increase of ≥50% over a 2-month period or Lymphocyte Doubling Time (LDT) in <6 months. LDT can be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months; patients with initial blood lymphocyte counts <30 × 109/L may require a longer observation period to determine the LDT. Factors contributing to lymphocytosis other than CLL (e.g., infections, steroid administration) should be excluded.
5. Autoimmune complications, including anaemia or thrombocytopenia poorly responsive to corticosteroids.
6. Symptomatic or functional extra-nodal involvement (e.g., skin, kidney, lung, spine).
7. Disease-related symptoms as defined by any of the following:

   1. Unintentional weight loss of ≥10% within the previous 06 months.
   2. Significant fatigue (i.e., ECOG performance scale 02 or worse; cannot work or unable to perform usual activities).
   3. Fever ≥100.5°F or 38.0°C for 02 or more weeks without evidence of infection.
   4. Night sweats for ≥1 month without evidence of infection.

   b. MCL Patients: i. Confirmed MCL with translocation t(11;14) (q13;q32) and/or overexpressed cyclin D1 ii. Measurable nodal disease (one or more lesions measuring ≥2 cm in the longest diameter) iii. Relapsed after, or were refractory to, 1-5 previous treatments

Exclusion Criteria:

1. Known prolymphocytic leukaemia, Central Nervous System (CNS) lymphoma or leukaemia; or known history of (or currently suspected) Richter's syndrome
2. Treatment with chemotherapy, external beam radiation therapy, anticancer antibodies, or investigational drug within 30 days of the first dose of study drug
3. Prior radio-conjugated or toxin-conjugated antibody therapy
4. Anticoagulation therapy (e.g., warfarin or equivalent vitamin K antagonists) within 07 days of the first dose of study drug.
5. Major surgery ≤30 days before the first dose of study drug
6. History of stroke or intracranial haemorrhage ≤6 months before the first dose of study drug
7. History of bleeding diathesis
8. Prior exposure to a B-cell lymphoma-2 (Bcl-2) inhibitor or B-cell receptor inhibitor like BTKs
9. Active Cytomegalovirus (CMV) infection or serologic status reflecting active Hepatitis B or C infection or known history of infection with Human Immunodeficiency Virus (HIV), or any uncontrolled active systemic infection.
10. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, Congestive Heart Failure, or Myocardial Infarction within 06 months of screening, or any Class 3 or 4 cardiac diseases as defined by the New York Heart Association Functional Classification, or QTcB >480 msec at screening.
11. Requiring treatment with proton-pump inhibitors (e.g., Omeprazole, Esomeprazole, Lansoprazole, Dexlansoprazole, Rabeprazole, or Pantoprazole).
12. Breastfeeding or pregnant.
13. Current life-threatening illness, medical condition, or organ/system dysfunction which, in the Investigator's opinion, could have compromised the subject's safety or put the study at risk.
14. Concurrent participation in another therapeutic clinical trial.

    -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- India (12):
  - Research Site, Ahmedabad
  - Research Site, Bangalore
  - Research Site, Bengaluru
  - Research Site, Chandigarh
  - Research Site, Gurugram
  - Research Site, Guwahati
  - Research Site, Hyderabad
  - Research Site, Kochi
  - Research Site, Kolkata
  - Research Site, Ludhiana
  - Research Site, Mumbai
  - Research Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220C00022&attachmentIdentifier=67c563ab-3e2b-42e6-a3a0-26b0d9ab3843&fileName=CSP_redacted.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220C00022&attachmentIdentifier=a374e585-97a1-447e-9e39-fed5d0570e96&fileName=SAP_redacted.pdf&versionIdentifier=
- See also: CSR_synopsis-redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8220C00022&attachmentIdentifier=7f653d0a-de43-48be-a693-3c29c9aa42b6&fileName=CSR_synopsis-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 participants were consented and were divided into two groups, participants with CLL/SLL (N=90) and participants with MCL (N=13). Out of these, 100 participants (89 in the CLL/SLL and 11 in the MCL group) were considered in the full analysis set, 03 enrolled participants were discontinued due to withdrawal of the consent form.
Groups:
- CCL/SLL: Participants were treatment naïve or had received at least one prior therapy
- Relapsed and Refractory MCL: Participants had received at least one prior therapy
Period: Overall Study
Arm/Group | CCL/SLL | Relapsed and Refractory MCL
Started | 90 | 13
Completed | 82 | 8
Not Completed | 8 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Disease Progression | 2 | 0
Not completed — Patient Decision | 4 | 2
Not completed — Death, Serious Adverse Event, Screen Failure | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCL/SLL | Relapsed and Refractory MCL | Total
Number analyzed (Participants) | 89 | 11 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (11.2) | 60.3 (6.9) | 61.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 2 | 20
  Male | 71 | 9 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 89 | 11 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Objective Response to Treatment
Description: The efficacy of acalabrutinib was assessed by measuring the participants' objective response to treatment.
  Objective response = Complete Response (CR) + Partial Response (PR) + Partial Response with lymphocytosis (PRL).
Time Frame: Visit 5 (Day 85) and Visit 8 (Day 170)
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- CLL/SLL: Participants were treatment naïve or had received at least one prior therapy
Arm/Group | CLL/SLL | Relapsed and Refractory MCL
Number analyzed (Participants) | 89 | 11
Participants
  Visit 5: CR | 1 | 2
  Visit 5: PR | 53 | 3
  Visit 5: PRL | 1 | 0
  Visit 5: Objective Response | 55 | 5
  Visit 8: CR | 4 | 0
  Visit 8: PR | 50 | 4
  Visit 8: PRL | 1 | 0
  Visit 8: Objective Response | 55 | 4

2. Primary Outcome: Adverse Events of Special Interest (AESI) Including Arrhythmias (Atrial Fibrillation), Anaemia, Hypertension, Bleeding, Infections
Description: The AESIs for acalabrutinib, including arrhythmias (atrial fibrillation), anaemia, hypertension, bleeding, and infections, are presented.
Time Frame: Throughout study completion, approximately 198 days (from the Screening Phase [Day 0], Treatment Phase [Days 1-170], and until the Follow-up Phase [28 days after Day 170])
Population: Safety Analysis Set
Measure: Number; unit: Events
Arm/Group | CLL/SLL | Relapsed and Refractory MCL
Number analyzed (Participants) | 89 | 11
Events | 0 | 0

3. Secondary Outcome: Health Related Quality of Life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 [EORTC QLQC30] Questionnaire)
Description: The EORTC QLQ-C30 is a 30-item questionnaire that measures quality of life in cancer patients. It is divided into several scales: Functioning Scales (Physical, Role, Cognitive, Emotional, and Social), Symptom Scales (Fatigue, Pain, Nausea/Vomiting), Dyspnoea, Sleep Disturbances, Appetite Loss, Diarrhoea, Constipation, Financial Difficulties, and Global Health Status/Quality of Life Scale. Scores range from 0 to 100. A higher score indicates better health related quality of life.
  The total scores were calculated from the mean of the 13 QLQ-C30 scales (Global Quality of Life Scale and Financial Impact Scale were excluded). Prior to calculating the mean, Symptom Scales were reversed to obtain a uniform direction of all scales. The total score was only calculated if all of the required 13 scale scores were available using scale scores based on the completed items, provided that at least 50% of the items in that scale were completed.
Time Frame: From Visit 1 (Day 0), during Visit 5 (Day 85), and at Visit 8 (Day 170)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | CLL/SLL | Relapsed and Refractory MCL
Number analyzed (Participants) | 89 | 11
Score on a scale
  Visit 1 Total Score | 56.9 (12.52) | 57.0 (6.46)
  Visit 5 Total Score | 56.8 (7.88) | 57.9 (7.21)
  Visit 8 Total Score | 57.9 (9.34) | 58.6 (6.76)

4. Primary Outcome: Second Primary Malignancies
Description: The safety of acalabrutinib was investigated by determining the number of second primary malignancies.
Time Frame: as for outcome 2
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | CLL/SLL | Relapsed and Refractory MCL
Number analyzed (Participants) | 89 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout study completion, approximately 198 days (from the Screening Phase [Day 0], Treatment Phase [Days 1-170], and until the Follow-up Phase [28 days after Day 170])
Arm/Group | CCL/SLL | Relapsed and Refractory MCL
All-Cause Mortality (participants affected / at risk) | 1/89 | 2/11
Serious Adverse Events (participants affected / at risk) | 8/89 | 3/11
Other Adverse Events (participants affected / at risk) | 38/89 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCL/SLL (N=89) | Relapsed and Refractory MCL (N=11)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CCL/SLL (N=89) | Relapsed and Refractory MCL (N=11)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (10) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (10) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Lipase (Investigations) | 1 (2) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovitaminosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Pallor (Vascular disorders) | 1 (2) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT04930536/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT04930536/SAP_001.pdf